CLINICAL TRIAL: NCT02322177
Title: Maternal Inborn Errors of Metabolism in Pregnancy: A Pregnancy Registry Protocol
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150049; 15-HG-0049
Record Dates: First submitted 2014-12-19; First posted 2014-12-23 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-09-09

CONDITIONS: Inborn Errors of Metabolism; Pregnancy; Acidemias
Keywords: Inborn Error of Metabolism; Pregnancy; Amino acid disorder; Fatty acid oxidation disorder; Organic Acidemia; Natural History
MeSH Terms: conditions — Metabolism, Inborn Errors; Amino Acid Metabolism, Inborn Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Participants are women with inborn errors of metabolism who have been pregnant

SUMMARY:
Background:

- People with inborn errors of metabolism can t turn food into energy the right way. This can affect a person s growth and health. Researchers want to know how this condition affects a pregnant woman and her baby.

Objectives:

- To collect data from the medical records of women with an inborn error of metabolism. Also, to create a pregnancy registry of inborn errors of metabolism.

Eligibility:

* Women with an inborn error of metabolism who either:
* have been pregnant in the past,
* are currently pregnant, or
* have recently talked with their doctor about becoming pregnant.

Design:

* This study will collect data only. No extra tests will be done.
* Participants will be in the study for the length of their pregnancy and for 1 year after delivery.
* Participants will answer questions about their family s health.
* The participant s doctor will send their medical records to researchers. These may include data about:
* Last health care visit before pregnancy
* Blood, urine, ultrasound, or lab results during pregnancy
* Delivery and recovery after delivery
* Researchers will ask for the test(s) used to confirm pregnancy.
* After the participant has her baby, researchers will ask for data about how the baby is doing. This may include when the baby is sitting, walking, talking, etc.
* The data will be placed into a database. The database will not include the participant s name or identifying data.

DETAILED DESCRIPTION:
Women with inherited metabolic disorders are reaching child bearing age more often due to advances in early diagnosis and improved pediatric care. For many of these disorders, there is very little information in the literature to guide the counseling and treatment of these patients and their pregnancies.

The most information for the effects of an underlying inborn error of metabolism in pregnancy derives from the study of phenylketonuria (PKU). From the knowledge gained through the collection of information from multiple cases of pregnancy affected by PKU, important management issues were identified. For example, children born to mothers with an unrestricted diet were substantially more likely to have intellectual disability, microcephaly, and low birth weights than women who maintained a phenylalanine restricted diet. The excess phenylalanine poses long-term health risks to the developing fetus and now a vigilant metabolic approach is recognized as mandatory in women with PKU desiring pregnancy.

Compared to PKU, most or all other intermediary metabolic disorders have been understudied. For example, there are nine published cases of methylmalonic acidemia (MMA) in pregnancy and one case of cobalamin C deficiency in pregnancy, and review articles have reported the same cases. For other inborn errors of metabolism there is even less published or known. The paucity of publication of pregnancy in IEMs other than PKU may be due to the lack of organized research to address pregnancy management in metabolic disorders.

The objective of this study is to establish a pregnancy registry of women with inborn errors of metabolism other than PKU. We will collect management plans, baseline laboratory values, prenatal and postpartum course including metabolic and obstetrical issues, and fetal/neonatal outcomes. This study will also investigate reproductive issues including infertility and use of artificial reproductive technologies. A registry of this type will allow physicians and patients to report varying management and outcomes, both positive and negative, with the broader goal of delineating optimal maternal and fetal outcomes for these unique patient populations. Our registry data would also serve as a vehicle to disseminate management experience for all providers, recognizing that individual centers may not have sufficient experience to make accurate management decisions on their own.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients clinically diagnosed with methylmalonic acidemia or another inborn error of metabolism are eligible to participate; mutational and enzymatic status is preferred but not required. Biochemical testing is required.
* Women with inborn errors of metabolism who have had a clinically documented prior pregnancy, currently are pregnant or planning a pregnancy.

EXCLUSION CRITERIA:

* Patients with phenylketonuria or hyperphenylalaninemia.
* Anyone unwilling to provide informed consent (for themselves as adults, or on behalf of their children as minors) or assent.
* Medical condition(s) or mental retardation are not in themselves reason for exclusion if in the judgment of the referring physician this would involve no more than minimal risk. We will make every effort to explain the study for the purpose of assent in a manner that the family feels is both age and developmentally appropriate for that child.
* We will review a clinical description from the referring physician about a potential research subject to determine that the subject is appropriate to enter into the study. We reserve the right to exclude cases that are not definitively diagnosed by metabolites and/or molecular genetics or related to our direct research interests. We expect this to be a rare minority.

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants are women with inborn errors of metabolism who have been pregnant
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2014-12-19; Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Maternal inborn errors of metabolism | Yearly

CONTACTS AND LOCATIONS:
Overall Officials: Charles P Venditti, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (2):
- United States (2):
  - National Human Genome Research Institute (NHGRI), Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

REFERENCES:
- [Background] Kuseyri O, Weissbach A, Bruggemann N, Klein C, Gizewska M, Karall D, Scholl-Burgi S, Romanowska H, Krzywinska-Zdeb E, Monavari AA, Knerr I, Yapici Z, Leuzzi V, Opladen T. Pregnancy management and outcome in patients with four different tetrahydrobiopterin disorders. J Inherit Metab Dis. 2018 Sep;41(5):849-863. doi: 10.1007/s10545-018-0169-0. Epub 2018 Mar 28. PMID 29594647
- [Background] Raval DB, Merideth M, Sloan JL, Braverman NE, Conway RL, Manoli I, Venditti CP. Methylmalonic acidemia (MMA) in pregnancy: a case series and literature review. J Inherit Metab Dis. 2015 Sep;38(5):839-46. doi: 10.1007/s10545-014-9802-8. Epub 2015 Jan 8. PMID 25567501
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-HG-0049.html